CLINICAL TRIAL: NCT02045446
Title: Maintenance Chemotherapy Versus Consolidative Stereotactic Body Radiation Therapy (SBRT) Plus Maintenance Chemotherapy for Stage IV Non-Small Cell Lung Cancer (NSCLC): A Randomized Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Puneeth Iyengar, ASSISTANT PROFESSOR, Radiation Oncology - RO-Radiation Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092013-070
Record Dates: First submitted 2014-01-14; First posted 2014-01-24 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Maintenance Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance chemotherapy (Active Comparator): FDA approved drugs for the study population: Bevacizumab, Docetaxel, Erlotinib, Gemcitabine, Pemetrexed
  Interventions: Drug: Maintenance chemotherapy
- Stereotactic Body Radiation Therapy (Experimental): consolidative Stereotactic Body Radiation Therapy (SBRT) plus maintenance chemotherapy
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Drug: Maintenance chemotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy
  Other Names: SBRT
  Arms: Stereotactic Body Radiation Therapy
Drug: Maintenance chemotherapy — Maintenance chemotherapy

SUMMARY:
The core hypothesis to be tested is that the use of consolidative SBRT followed by maintenance chemotherapy in patients with less than or equal to 6 metastatic sites (primary + 5) will improve progression free survival (PFS) compared to maintenance chemotherapy alone.

DETAILED DESCRIPTION:
This protocol is a randomized phase II trial of maintenance chemotherapy versus consolidative Stereotactic Body Radiation Therapy (SBRT) plus maintenance chemotherapy for patients with Stage IV non-small cell lung cancer (NSCLC).

Prior to accrual on the trial, patients with Stage IV NSCLC will be treated with standard first-line chemotherapy. Patients who achieve a partial response or stable disease by imaging criteria with fewer than or equal to six sites of oligometastatic disease will be randomized to maintenance chemotherapy or consolidative SBRT to all sites of disease (followed by maintenance chemotherapy at the medical oncologist's discretion). Choices of first line and maintenance chemotherapy will be determined by the medical oncologist based on clinical appropriateness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy proven metastatic NSCLC (Stage IV).
2. Patients must have received first line chemotherapy, from 4-6 cycles, and achieved stable disease or a partial response.
3. Patients receiving first-line erlotinib, crizotinib for EGFR mutant-positive or EML4-ALK positive NSCLC will be excluded.
4. Age ≥ 18 years
5. Patients must have measurable disease at baseline.
6. Patients can have up to only 6 discrete active extracranial lesions (≤3 in the liver and ≤3 in the lung) identified by diagnostic CT or PET/CT scan or MRI within 8 weeks prior to the initiation of SBRT.

   1. For patients who have received prior radiotherapy to the primary site in the lung, residual PET activity is difficult to interpret and will not be considered a site of active disease if the CT appearance is stable or improved over an interval of at least three months
   2. Patients who previously received radiotherapy to the primary site will be ineligible if there is CT evidence of disease progression within the past 3 months.
   3. Patients with previously un-irradiated primary sites will be potentially eligible, but special considerations apply (section 4.3.2).
   4. Up to 2 contiguous vertebral metastases will be considered a single site of disease.
7. Patients must have a KPS >60
8. AST, ALT & Alkaline phosphates must be ≤ 2.5X the upper limit of normal. Total bilirubin must be within the limit of normal.
9. Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm³.
10. Patients should have adequate renal function (serum creatinine ≤1.5 times the ULN).
11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    11.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
12. Patients who would be receiving SBRT for lung tumors who are known or suspected by the treating radiation oncologist to have compromised lung function must have a documented forced expiratory volume in 1 second (FEV1) ≥ 1L.
13. Patients must provide verbal and written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who previously received radiotherapy to the primary site with CT evidence of disease progression at the primary site within 3 months following the initial radiotherapy.
2. Patients with untreated brain metastases Patients with serious, uncontrolled, concurrent infection(s).
3. Significant weight loss (>10%) in the prior 3 months.
4. Because the tolerance dose of SBRT to the gastrointestinal tract is not established, patients with metastatic disease invading the esophagus, stomach, intestines, or mesenteric lymph nodes will not be eligible.
5. Patients with cutaneous metastasis of NSCLC.
6. Patients with more than 6 discrete extra-cranial lesions.
7. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
8. Unwillingness to participate or inability to comply with the protocol for the duration of the study.
9. Patients who are pregnant. Patients with reproductive capability will need to use adequate contraception during the time of participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puneeth Iyengar, MD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiation Therapy: Consolidative Stereotactic Body Radiation Therapy (SBRT) plus maintenance chemotherapy
  Stereotactic Body Radiation Therapy
  Maintenance chemotherapy: Maintenance chemotherapy
Period: Overall Study
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Customized [Median (Full Range); unit: years]
  Age | 70.0 [51.0 to 79.0] | 63.5 [50.0 to 78.0] | 66 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 11 | 9 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29
Histology [Count of Participants; unit: Participants]
  Squamous | 3 | 1 | 4
  Nonsquamous | 12 | 13 | 25
Sites of disease prior to induction chemotherapy [Median (Full Range); unit: sites of disease] | 2 [2 to 5] | 3 [2 to 6] | 3 [2 to 6]
Previously treated brain metastases [Count of Participants; unit: Participants]
  Yes | 5 | 6 | 11
  No | 10 | 8 | 18
Induction chemotherapy, median cycles [Median (Full Range); unit: cycles] | 4 [4 to 6] | 4.5 [4 to 6] | 4 [4 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Evaluate the effect of SBRT with maintenance chemotherapy versus maintenance chemotherapy alone on progression free survival. Time to the development of new lesions, progression of existing lesions, or death, whichever came first, represented the primary end point of progression-free survival. All evaluations of disease response used RECIST (v1.1) criteria, in which progressive disease is defined as "At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm."
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15 | 14
months | 3.5 [3.387 to 4.315] | 9.7 [9.587 to 10.515]
Statistical Analysis 1: Comparison: Maintenance Chemotherapy vs Stereotactic Body Radiation Therapy; Test type: Superiority; p = .01, Log Rank; Hazard Ratio (HR) = .304, 95% CI 2-sided [0.113 to 0.815]

2. Secondary Outcome: In-field Local Control Versus Out-of-field Disease Progression
Description: Number of occurances of in-field local control and rate of out-of-field disease progression
Time Frame: 5 years
Measure: Number; unit: Patients
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15 | 14
Patients
  Progression in brain | 4 | 1
  Progression in liver | 0 | 2
  Progression in lung | 8 | 0
  Progression in bone | 1 | 1
  Progression in pancreas | 0 | 1
  In-field progression | 7 | 0

3. Secondary Outcome: Toxicities
Description: To evaluate the safety of SBRT with metastatic NSCLC after prior chemotherapy
Time Frame: 2 years
Measure: Number; unit: adverse events
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15 | 14
adverse events
  Grade 3 toxicities probably or definitely attributed to study | 2 | 4
  Grade 4 toxicities probably or definitely attributed to study | 1 | 0
  Grade 5 toxicities probably or definitely attributed to study | 0 | 0

4. Secondary Outcome: Overall Survival
Description: To evaluate overall survival after SBRT followed by maintenance chemotherapy in comparison to maintenance chemotherapy alone.
Time Frame: 5 years
Measure: Median (Full Range); unit: days
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15 | 14
days | 189 [28 to 587] | 203.5 [5 to 679]

5. Secondary Outcome: Duration of Maintenance Chemotherapy
Description: To evaluate the duration of maintenance chemotherapy and time to initiation of third line systemic agent (chemotherapy or biologic agent)
Time Frame: 5 years
Measure: Median (Full Range); unit: cycles
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 15 | 14
cycles | 3 [1 to 15] | 5 [3 to 19]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Maintenance Chemotherapy | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 3/15 | 3/14
Serious Adverse Events (participants affected / at risk) | 6/15 | 8/14
Other Adverse Events (participants affected / at risk) | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Chemotherapy (N=15) | Stereotactic Body Radiation Therapy (N=14)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Headaches (General disorders) | 1 (3) | 0 (0)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 0 (0) | 2 (3)
White blood cell count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Chemotherapy (N=15) | Stereotactic Body Radiation Therapy (N=14)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergy (seasonal) (Immune system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (4) | 3 (4)
Chills (General disorders) | 3 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 11 (16)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 4 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Dysesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (15)
Edema (General disorders) | 2 (2) | 2 (3)
Edema limbs (General disorders) | 3 (3) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Erythema multitforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Fatigue (General disorders) | 13 (17) | 8 (13)
Fever (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Shingles (Immune system disorders) | 1 (1) | 0 (0)
Oral lesions (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Low white blood count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 3 (3)
Lymphocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (10)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (6) | 5 (8)
Parathesia (tingling) (Nervous system disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Weakness (facial) (General disorders) | 1 (1) | 0 (0)
Weakness (limb) (General disorders) | 2 (2) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Bone marrow biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Throat pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dementia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT02045446/Prot_SAP_002.pdf